CLINICAL TRIAL: NCT03781128
Title: Safety and Efficacy of Lysergic Acid Diethylamide (LSD) as Treatment for Cluster Headache: a Randomized, Double-blind, Placebo-controlled Phase II Study
Brief Title: Lysergic Acid Diethylamide (LSD) as Treatment for Cluster Headache
Acronym: LCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC 2018-01082
Record Dates: First submitted 2018-11-07; First posted 2018-12-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cluster Headache
Keywords: lysergic acid diethylamide (LSD); serotonin; hallucinogen; cluster headache
MeSH Terms: conditions — Cluster Headache | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled two-phase cross-over study design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSD, Placebo (Other): Lysergic acid diethylamide (3 x 100 µg LSD in three weeks, per os) followed by Placebo
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: Placebo
- Placebo, LSD (Other): Placebo (3 x 1 vial looking like LSD in three weeks, per os) followed by Lysergic acid diethylamide
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: Placebo

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide — 100 µg, per os, 3 times within 3 weeks
  Other Names: LSD
Drug: Placebo — placebo in an identical-looking vial as LSD, per os, 3 times within 3 weeks

SUMMARY:
Background: After no official research in humans in the last 40 years, research and therapeutic uses of the serotonergic psychedelic lysergic acid diethylamide (LSD) are now re-recognized and include its use in brain research, alcoholism, anxiety associated with terminal illness, and treatment of headache disorders. Specifically, LSD has been reported to abort attacks, to decrease frequency and intensity of attacks, and to induce remission in patients suffering from cluster headache (CH).

Objective: To investigate the effects of an oral LSD pulse regimen (3 x 100 µg LSD in three weeks) in patients suffering from CH compared with placebo.

Design: Double-blind, randomized, placebo-controlled two-phase cross-over study design.

Participants: 30 patients aged ≥ 25 and ≤ 75 years with chronic or episodic CH with predictable periods lasting approximately 2 months and attacks responding to oxygen.

Main outcome measures: Changes in frequency and intensity of CH attacks assessed with a standardized headache diary Significance: CH is often rated as the most painful of all primary headaches, which not only causes significant disability, but is also associated with enormous personal, economic, and psychiatric burden. At the moment, there is no specific treatment available for CH, but serotonergic compounds represent an important drug class, especially in the abortive management of cluster attacks. However, there is a need for new treatment approaches, as CH is also often insufficiently managed with available medication. This study will evaluate the potential benefit and safety of a treatment with LSD for patients with CH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 25 and ≤ 75 years
* Chronic cluster headache (according to the International Headache Society (IHS) criteria) OR
* Episodic cluster headache (according to the IHS criteria) with recurrent predictable episodes lasting approximately 2 months and expected ongoing cluster period for at least one month beyond the inclusion
* Attacks respond to oxygen
* Sufficient understanding of the study procedures and risks associated with the study
* Participants must be willing to adhere to the study procedures and sign the consent form
* Participants are willing to abstain from taking preventive and abortive medication (except from oxygen) long enough before and after the LSD/placebo treatment session to avoid the possibility of a drug-drug interaction
* Participants are willing to refrain from taking any psychiatric medications during the experimental session period. If they are being treated with antidepressants, lithium or are taking anxiolytic medications on a fixed daily regimen, such drugs must be discontinued long enough before the LSD/placebo treatment session to avoid the possibility of a drug-drug interaction.
* Participants must also refrain from the use of any psychoactive drugs and caffeine within 24 hours of each LSD/placebo treatment session. They must agree not to use nicotine for at least 2 hours before and 6 hours after each dose of LSD. They must agree to not ingest alcohol-containing beverages for at least 1 day before each LSD treatment session. Non-routine medications for treating breakthrough pain taken in the 24 hours before the LSD treatment session may result in rescheduling the treatment session to another date, with the decision at the discretion of the investigators after discussion with the participant.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 24 hours after LSD/placebo administration.

Exclusion Criteria:

* Other forms of headache attacks (migraine, paroxysmal hemicranias, shortlasting unilateral neuralgiform headache attacks with conjunctival injection, tearing, sweating and rhinorrhea (SUNCT) or with cranial autonomic symptoms (SUNA))
* Women who are pregnant, nursing or of child-bearing potential and are not practicing an effective means of birth control (double-barrier method, i.e. pill/intrauterine device and preservative/diaphragm)
* Past or present diagnosis of a primary psychotic disorder. Subjects with a first degree relative with psychotic disorders are also excluded.
* Past or present bipolar disorder (DSM-IV).
* Current substance use disorder (within the last 2 months, DSM-V, except nicotine).
* Somatic disorders including severe cardiovascular disease, untreated hypertension (systolic blood pressure > 160mmHg without treatment, systolic blood pressure > 140 mmHg with treatment), severe liver disease (liver enzymes increase by more than 5 times the upper limit of normal) or severely impaired renal function (estimated creatinine clearance <30 ml/min), or other that in the judgement of the investigators pose too great potential for side effects.
* Weight < 45kg
* Participation in another clinical trial (currently or within the last 30 days)
* Participants taking higher steroid doses (>10mg/d) over a longer time period (>2 weeks), as this would require tapering
* Use of immunomodulatory agents (i.e. azathioprine) in the past 2 weeks
* Use of serotonergic antiemetics (i.e. ondansetron) in the past 2 weeks

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of the cluster headache attacks | 8 weeks before and after pulse regimen
  assessed with a standardized headache diary, within-subjects analysis
Change in intensity of the cluster headache attacks | 8 weeks before and after pulse regimen
  assessed with a standardized headache diary, within-subjects analysis

SECONDARY OUTCOMES:
Episode abortion | through study completion, an average of 1 year
  assessed with a standardized headache diary
Change in duration of attacks | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Time to first attack after completion of pulse regimen | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Cumulative time with headache | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Change in cluster period duration and interval between cluster periods | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Number of attacks requiring abortive medication | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Number of Attack-associated autonomic symptoms | 8 weeks after pulse regimen
  assessed with a standardized headache diary
Quality of life assessed by questionnaires: 36-item short-form health survey (SF-36) | through study completion, an average of 1 year
  assessment with the validated 36-item short-form health survey (SF-36), which measures health-related quality of life
Quality of life assessed by questionnaires: 5-level EuroQoL-5D (EQ-5D-5L) | through study completion, an average of 1 year
  assessment with the 5-level EuroQoL-5D (EQ-5D-5L), which is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life
Quality of life assessed by questionnaires: Headache Impact Test (HIT-6) | through study completion, an average of 1 year
  assessment with the Headache Impact Test (HIT-6), which measures the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning and psychological distress.
Effects on depressive /anxious symptoms assessed by questionnaires: State-trait anxiety inventory (STAI) | through study completion, an average of 1 year
  assessment with the State-trait anxiety inventory (STAI), which measures anxiety
Effects on depressive /anxious symptoms assessed by questionnaires: Generalized anxiety disorder-7 (GAD-7) | through study completion, an average of 1 year
  assessment with the Generalized anxiety disorder (GAD-7), which measures anxiety
Effects on depressive /anxious symptoms assessed by questionnaires: Hospital Anxiety and Depression Scale (HADS) | through study completion, an average of 1 year
  assessment with the Hospital Anxiety and Depression Scale (HADS), which measures anxiety and depression severity
Effects on depressive /anxious symptoms assessed by questionnaires: Beck Depression Inventory (BDI) | through study completion, an average of 1 year
  assessment with the Beck Depression Inventory (BDI), which measures depression
Effects on depressive /anxious symptoms assessed by questionnaires: Patient health questionnaire-9 (PHQ-9) | through study completion, an average of 1 year
  assessment with the Patient health questionnaire-9 (PHQ-9), which measures depression
Acute autonomic effects assessed by blood pressure | 10 hours after drug administration
  systolic and diastolic blood pressure in mmHg
Acute autonomic effects assessed by heart rate | 10 hours after drug administration
  heart rate in beats per minute
Acute autonomic effects assessed by body temperature | 10 hours after drug administration
  body temperature in °Celsius
Adverse Events | through study completion, an average of 1 year
  adverse events will be recorded
Acute psychological effects assessed by questionnaire Visual analogue scales (VAS) | 10 hours after drug administration
  assessment of subjective effects using visual analogue scales
Acute psychological effects assessed by SCQ | 10 hours after drug administration
  assessed with the states of consciousness questionnaire (SCQ)
Acute psychological effects assessed by questionnaire 5-dimensions of altered states of consciousness | 10 hours after drug administration
  assessed with the 5-dimensions of altered states of consciousness questionnaire (5D-ASC)
Persisting effects attributed to the LSD experience | through study completion, an average of 1 year
  assessment of persisting effects with the persisting effects questionnaire (PEQ) which assesses changes in attitude, mood, behavior and spiritual experience. The questionnaire will be completed at the beginning, after pulse regimens, and at the end of the study.
Change of attack frequency at the end of the study compared with baseline | through study completion, an average of 1 year
  pre-post study comparison in all subjects, assessed with a standardized headache diary
Change of attack intensity at the end of the study compared with baseline | through study completion, an average of 1 year
  pre-post study comparison in all subjects, assessed with a standardized headache diary
Change in attack frequency before and after pulse regimen | 8 weeks after first pulse regimen
  between-subjects analysis before cross-over, assessed with a standardized headache diary
Change in attack intensity before and after pulse regimen | 8 weeks after first pulse regimen
  between-subjects analysis before cross-over, assessed with a standardized headache diary
Blinding | after study days and at the end of study visit
  patients and investigators will be asked at the end of a study day and and the end of the study visit to guess the drug treatment
Expectancy | at screening
  a modified 2-item version of the Credibility / Expectancy Questionnaire (CEQ) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Liechti, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No